CLINICAL TRIAL: NCT06631612
Title: Daily Versus Alternate Day Regimen of Iron Supplementation in Children with Iron Deficiency Anemia: a Hospital Based Study
Brief Title: Daily Versus Alternate Day Regimen of Iron Supplementation in Children with Iron Deficiency Anemia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omnya atef Mahmoud Abdelbaky, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD288/2023
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Iron Deficiency Anemia Treatment
Keywords: iron defiiency; Anemia; hepcidin
MeSH Terms: conditions — Anemia | interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- daily dose of Iron Supplementation (Active Comparator): daily dose of 3 mg/kg elemental Iron before bed
  Interventions: Drug: ferric hydroxide polymaltose complex; Drug: Albendazole.
- alternate day regimen (Experimental): every other day dose of 3mg/kg elemental Iron before bed
  Interventions: Drug: ferric hydroxide polymaltose complex; Drug: Albendazole.

INTERVENTIONS:
Drug: ferric hydroxide polymaltose complex — participants will receive oral iron supplementation according to body weight every other day
  Arms: alternate day regimen
Drug: ferric hydroxide polymaltose complex — participants will receive oral iron supplementation dose according to body weight daily
  Arms: daily dose of Iron Supplementation
Drug: Albendazole. — both arms will receive Albendazole 400mg once at the beginning f the study to be repeated after 1 week

SUMMARY:
The goal of this clinical trial is to learn if giving iron supplementation every other day is as effective as giving it daily in children with Iron Deficiency Anemia.

The main questions it aims to answer are:

1. Will alternate day regimen improve hemoglobin and iron profile just as well as daily dose?
2. Which group will suffer less side effects from Iron Supplementation?

Participants will be divided into two groups:

Group A: will receive oral Iron supplementation daily for 2 months Group B: will receive oral Iron supplementation every other day for 2 months Participants will be monitored using weekly phone calls to insure compliance and report side effects.

Both groups will be given Albendazole 400 mg once at the beginning of the study to be repeated in 1 week

DETAILED DESCRIPTION:
Children will be recruited from the pediatrics general clinic in Al Demerdash Hospital.

After checking fro inclusion and exclusion criteria and signing the informed consent form the following will be carried out.

1-History taking: Caregivers will be asked about:

1. Sociodemographic data: using a self-structured questionnaire

   * Age of the child
   * Gender of the child
   * Order of birth
   * Consanguinity
   * Mode of delivery (either vaginal delivery or by c-section)
   * Age of the mother and father
   * Level of education or the mother and father
   * Address of the family
2. Questions about risk factors for iron deficiency anemia/ to exclude other causes of anemia:

   * Prematurity / low birth weight.
   * Duration of exclusive breast feeding
   * Consumption of cow milk before 1 year of age/excessive consumption of cow milk
   * Mother's iron status during pregnancy
   * family history for hemolytic anemias or regular blood transfusions.
   * history of blood transfusions (or hemolysis: pallor ,jaundice, dark urine,anemia)
   * History of chronic illness (Cardiac, hepatic or renal patients).
   * History of chronic blood loss
3. Questions about symptoms of iron deficiency anemia:

Headache, lack of concentration,fatigue, palpitations, irritability,fainting, wanting to eat odd substances such as dirt or ice (also called pica),,,,etc.

2-Examination:

General examination:

1. Anthropometric measures (weight,height,BMI).
2. Look for signs of anemia: Pallor, brittle hair and nails,angular stomatitis,glossitis, Koilonychia or spooning of nails, tachycardia, hyperdynamic circulation.
3. Abdominal examination: look for tenderness, masses or hepatosplenomegaly. 3-Investigations: (a blood sample of about 5 ml will be drawn twice, once at presentation and again after 8 weeks) Complete Blood Picture (CBC) Iron profile: serum iron, TIBC. Participants will be divided into two groups.

Both groups will receive:

1. Health education regarding IDA including:

   Prenatal and postnatal nutrition, the definition of anemia, diagnosis of anemia, factors causing anemia, sources of heme and non-heme iron, foods and nutrients that interfere with and promote iron absorption, and the impact of anemia on toddlers. Also food sources high in nutrients and processing high iron content of complementary breastfeeding.
2. Treatment for parasitic infections (deworming ) Albendazole 400 mg once.

Then:

Group (1) will receive daily dose of 3 mg/kg ferrous fumarate before bed. Group (2) will receive a dose of 6mg/kg ferrous fumarate before bed every other day with a maximum dose of 180 mg /day.

Participants will be dedicated to the study for 8 weeks. During this time, they will be monitored using weekly phone calls to:

1. Reinforce the health education message.
2. make sure they are compliant to their treatment.
3. monitor if any new symptoms or side effects appear.

   * Outcomes:

Participants will be followed for 8 weeks. Check in after 8 weeks to repeat hemoglobin levels and serum Iron and TIBC.

ELIGIBILITY:
Inclusion Criteria:

children 2-12 years of age diagnosed wit Iron Deficiency anemia according to WHO criteria (hemoglobin below 11 g/dl and transferrin saturation below 16%)

Exclusion Criteria:

1. Children already being treated for iron deficiency anemia
2. Children known to have hemolytic anemias
3. Children with GIT disorders that prevent iron absorption (Inflammatory bowel disease,celiac disease …etc)
4. Children with chronic diseases (heart disease,liver disease,kidney disease, endocrinological disease).
5. Children who are underweight or morbidly obese

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
change in hemoglobin | 8 weeks
  treatment will be considered successful if there is an increase of hemoglobin at least 1 g/dl every 4 weeks
change in Iron Profile | 8 weeks
  changes in serum Iron will be compared between the two groups
change in iron profile | 8 weeks
  change in TIBC will be compared between the two groups
change in iron profile | 8 weeks
  change in transferrin saturation will be compared between the two groups

SECONDARY OUTCOMES:
frequency of side effects | 8 weeks
  frequency of different side effects (eg: abdominal pain, nausea, vomitting , etc.)will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Wessam A Professor, MD, Study Director — Ain Shams Pediatrics Hospital
Locations (1):
- Ain Shams University Hospitals, Cairo, Abaseya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data collected and used in the results will be shared
Supporting Information: Study Protocol, SAP
Time Frame: start date: June 2025 end date: June 2026
Access Criteria: Anyone can access the IPD plan including the excel sheet of data collection and what type of analysis was used.
URL: https://osf.io/